CLINICAL TRIAL: NCT06154109
Title: Comparative Efficacy of Xiaopi Granules and Decoction in Improving Pathological Complete Response of Neoadjuvant Chemotherapy of Triple-negative Breast Cancer: a Randomized, Double-blind, Controlled Trial
Brief Title: Comparative Efficacy of Xiaopi Granules and Decoction in Triple-negative Breast Cancer: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhiyu Wang (Other)
Responsible Party: Sponsor-Investigator, Zhiyu Wang, professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Organization: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GuangdongXPRCT
Record Dates: First submitted 2023-10-31; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Triple Negative Breast Neoplasms
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Xiaopi granules plus neoadjuvant chemotherapy (Experimental): Xiaopi granules have a dosage of 18 g per bag, 18 g per administration, twice daily, for a total of 8 days per treatment course. The duration of the treatment course will align with that of the chemotherapy regimen. The neoadjuvant chemotherapy is developed based on the National Comprehensive Cancer Network (NCCN) guidelines. Different treatments and doses are according to the standard recommendations outlined in the guidelines. Treatment options may include AC-T, ECT, EC, TC, AC, TAC, TP, etc.
  Interventions: Drug: Xiaopi granules
- Xiaopi decoction plus neoadjuvant chemotherapy (Experimental): Xiaopi decoction has a dosage of 18 g per bag, 18 g per administration, twice daily, for a total of 8 days per treatment course. The duration of the treatment course will align with that of the chemotherapy regimen. The neoadjuvant chemotherapy is developed based on the National Comprehensive Cancer Network (NCCN) guidelines. Different treatments and doses are according to the standard recommendations outlined in the guidelines. Treatment options may include AC-T, ECT, EC, TC, AC, TAC, TP, etc.
  Interventions: Drug: Xiaopi decoction
- Placebo plus neoadjuvant chemotherapy (Placebo Comparator): The placebo is a look-alike substance that contains no active drug and has a placebo inspection report. The dosage of 18g per bag, 18g per administration, twice daily, for a total of 8 days per treatment course. The duration of the treatment course will align with that of the chemotherapy regimen. The neoadjuvant chemotherapy is developed based on the National Comprehensive Cancer Network (NCCN) guidelines. Different treatments and doses are according to the standard recommendations outlined in the guidelines. Treatment options may include AC-T, ECT, EC, TC, AC, TAC, TP, etc.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xiaopi granules — Xiaopi granules (18 g/ bag), 18 g/ time, 2 times/day, 8 days/course.
  Other Names: Xiaopi formula
  Arms: Xiaopi granules plus neoadjuvant chemotherapy
Drug: Xiaopi decoction — Xiaopi decoction (18 g/ bag), 18 g/ time, 2 times/day, 8 days/course.
  Other Names: Xiaopi formula
  Arms: Xiaopi decoction plus neoadjuvant chemotherapy
Drug: Placebo — The placebo does not contain any active pharmaceutical ingredients .
  Arms: Placebo plus neoadjuvant chemotherapy

SUMMARY:
The goal of this clinical trial is to compare the efficacy of xiaopi granules and decoction in improving the pathological complete response (pCR) of neoadjuvant chemotherapy of triple-negative breast cancer. The main objective aims to answer whether Xiaopi granules combined with neoadjuvant Chemotherapy could improve the pCR rate of triple-negative breast cancer. The secondary outcome included genomics of plasma extracellular vesicles, plasma metabolites and metabolomics, urine metabolomics, fecal intestinal flora tests, pathological tissue genomics, functional assessment of cancer therapy breast (FACT-B), and adverse events.

Participants enrolled in this study will be randomized to xiaopi granules plus neoadjuvant chemotherapy, or xiaopi decoction plus neoadjuvant chemotherapy, or placebo plus neoadjuvant chemotherapy alone.

Researchers will compare the pathological complete response between xiaopi granules and decoction group, and to determine their effects in chemosensitizing triple-negative breast cancer.

DETAILED DESCRIPTION:
Background: Triple-negative breast cancers (TNBCs) are characterized by poor prognosis, rapid progression to metastatic stage, and onset of resistance to chemotherapy. Neoadjuvant chemotherapy is commonly used to improve the surgical pathological complete response rate (pCR) in stage II-III triple-negative breast cancer. However, chemotherapy can lead to immune escape and drug resistance in breast cancer cells, while the toxic side effects significantly affect patients' quality of life. The combination of Chinese herbal medicine and chemotherapy can improve survival rates while alleviating chemotherapy-related adverse events. Xiaopi Granules were developed by Professor Lin Yi, a renowned Traditional Chinese Medicine doctor in the field of breast diseases. The investigators' preliminary research has confirmed that Xiaopi Granules can inhibit tumor progression by targeting TAMs/CXCL1 signaling to suppress chemotherapy-induced autophagy, as well as inhibit the formation of tumor stem cells and pre-metastatic niches. Chinese medicine granules not only have several advantages compared to decoction, such as reliable drug quality and convenient administration but also have the characteristics of individualized prescription. However, whether their efficacy is comparable to that of the decoction granules still requires exploration. The investigators aimed to compare the efficacy of xiaopi granules and decoction in improving the pathological complete response of neoadjuvant chemotherapy of triple-negative breast cancer.

Hypothesis: Xiaopi granules can improve the pathological complete response of neoadjuvant chemotherapy of triple-negative breast cancer.

Patients and methods: Ninety patients with TNBC will be enrolled in this study and randomized to xiaopi granules plus neoadjuvant chemotherapy, xiaopi decoction plus neoadjuvant chemotherapy, or placebo plus neoadjuvant chemotherapy. The primary aim is the rate of pathological complete response (pCR, defined as the absence of invasive cells in breast and lymph nodes). The secondary outcome included genomics of plasma extracellular vesicles, plasma metabolites and metabolomics, urine metabolomics, fecal intestinal flora tests, pathological tissue genomics, functional assessment of cancer Therapy-Breast(FACT-B), and safety( AE and SAE). The neoadjuvant chemotherapy is carried out based on the National Comprehensive Cancer Network (NCCN) guidelines. Different treatments and doses are set according to the standard recommendations outlined in the guidelines. In addition to receiving neoadjuvant chemotherapy, the participants will be subjected to Xiaopi granules or decoction orally at a dosage of 18g per bag, twice daily, for a total of 8 days per treatment course. The duration of the treatment course will align with that of the chemotherapy regimen. A placebo is a look-alike substance that contains no active drug.

ELIGIBILITY:
Inclusion Criteria:

* Females aged ≥18 and ≤75 years
* Pathological diagnosis of triple-negative breast cancer with stage II-III
* Not having received any previous treatment for breast cancer
* Having at least one measurable tumor
* No distant metastases
* ECOG score 0-2
* Neoadjuvant chemotherapy or combination immunotherapy
* Agree to participate in this clinical study and sign the informed consent form

Exclusion Criteria:

* Pregnant and breastfeeding, with fertility requirements during the study period
* Combined other malignant tumors
* Combination of serious diseases of the heart, brain, liver, kidney, and hematopoietic system, liver function impairment, and diabetes mellitus
* Active hepatitis B virus or hepatitis C virus infection, or human immunodeficiency virus (HIV) infection
* Presence of factors affecting the administration and absorption of the drug
* Allergy to the drug components of this regimen
* A history of psychotropic substance abuse or drug use
* The patient has other life-threatening diseases
* Participating in other drug trials

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-25 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | Through study completion,an average of 6 moths
  Defined as the absence of invasive cells in breast and lymph nodes.

SECONDARY OUTCOMES:
Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Through study completion, an average of 6 moths
  The RECIST 1.1 version is used as the standard for evaluating the clinical efficacy of solid tumors.
Genomics of plasma extracellular vesicles | Through study completion, an average of 6 moths
  Extracellular vesicles were isolated from the plasma of breast cancer patients using a differential ultracentrifugation method. High-throughput whole transcriptome sequencing was conducted to identify differentially expressed genes in the isolated extracellular vesicles. The primary experimental procedures for transcriptome sequencing analysis include RNA quantification and qualification, library preparation for transcriptome sequencing, clustering and sequencing, and data analysis. . Analysis of whole transcriptome microarray data was performed using BioConductor software based on the statistical R programming language.
Plasma Genomic Tests | Through study completion, an average of 6 moths
  Utilize the Ultimate U3000 HPLC (Thermo Fisher Scientific) coupled to Q Exactive Plus mass spec- trometer (Thermo Fisher Scientific) to detect differences in metabolites within the blood of different medication intervention treatment groups before and after medication.All data were acquired and analyzed with the Xcalibur 4.0 software (Thermo Fisher Scientific).
Urine Metabolomics Tests | Through study completion, an average of 6 moths
  Utilize the Vanquish ultra-high-performance liquid chromatography-mass spectrometry system (Thermo Fisher Scientific) to detect variations in metabolites within the urine of different medication intervention treatment groups before and after medication.All data were acquired and analyzed with the Xcalibur 4.0 software (Thermo Fisher Scientific).
Fecal Intestinal Flora Tests | Through study completion, an average of 6 moths
  Laboratory testing for differences in faecal intestinal flora testing before and after the patient's medication.
Pathological Tissue Genomics Tests | Through study completion, an average of 6 moths
  Using whole exome sequencing (WES) to perform high-throughput sequencing of the exonic regions in pathological tissues, thereby detecting mutations, insertions, or deletions within genes. Furthermore, utilize the Genome Analysis Toolkit (GATK) software package to analyze the genomic sequencing data.
Functional Assessment of Cancer Therapy-Breast | Through study completion, an average of 6 moths
  Utilize the FACT-B questionnaire to evaluate the quality of life of breast cancer patients in different medication intervention treatment groups before and after treatment. This questionnaire comprehensively assesses patients' performance in social interactions, emotional experiences, daily functioning, and physical condition, which indirectly reflects their overall quality of life.
Safety assessments | Through study completion, an average of 6 moths
  Evaluate to adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyu Wang, PhD, Study Chair — Guangdong Provincial Hospital of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No
Firstly, sharing IPD could potentially lead to the identification of individual participants, breaching their privacy rights. It is crucial to prioritize the protection of personal information and ensure that participants' identities remain confidential. Secondly, participants trust that their data will be used responsibly and for the intended purpose of the study. Sharing IPD without their explicit consent may go against ethical guidelines and compromise the trust between researchers and participants.

REFERENCES:
- [Background] Foulkes WD, Smith IE, Reis-Filho JS. Triple-negative breast cancer. N Engl J Med. 2010 Nov 11;363(20):1938-48. doi: 10.1056/NEJMra1001389. PMID 21067385
- [Background] Nedeljkovic M, Damjanovic A. Mechanisms of Chemotherapy Resistance in Triple-Negative Breast Cancer-How We Can Rise to the Challenge. Cells. 2019 Aug 22;8(9):957. doi: 10.3390/cells8090957. PMID 31443516
- [Background] Park YH, Lal S, Lee JE, Choi YL, Wen J, Ram S, Ding Y, Lee SH, Powell E, Lee SK, Yu JH, Ching KA, Nam JY, Kim SW, Nam SJ, Kim JY, Cho SY, Park S, Kim J, Hwang S, Kim YJ, Bonato V, Fernandez D, Deng S, Wang S, Shin H, Kang ES, Park WY, Rejto PA, Bienkowska J, Kan Z. Chemotherapy induces dynamic immune responses in breast cancers that impact treatment outcome. Nat Commun. 2020 Dec 2;11(1):6175. doi: 10.1038/s41467-020-19933-0. PMID 33268821
- [Background] Mehraj U, Dar AH, Wani NA, Mir MA. Tumor microenvironment promotes breast cancer chemoresistance. Cancer Chemother Pharmacol. 2021 Feb;87(2):147-158. doi: 10.1007/s00280-020-04222-w. Epub 2021 Jan 9. PMID 33420940
- [Background] Shree T, Olson OC, Elie BT, Kester JC, Garfall AL, Simpson K, Bell-McGuinn KM, Zabor EC, Brogi E, Joyce JA. Macrophages and cathepsin proteases blunt chemotherapeutic response in breast cancer. Genes Dev. 2011 Dec 1;25(23):2465-79. doi: 10.1101/gad.180331.111. PMID 22156207
- [Background] Shi G, Yu D, Wu J, Liu Y, Huang R, Zhang CS. A systematic review and meta-analysis of traditional Chinese medicine with chemotherapy in breast cancer. Gland Surg. 2021 May;10(5):1744-1755. doi: 10.21037/gs-21-284. PMID 34164318
- [Background] Wang S, Liu X, Huang R, Zheng Y, Wang N, Yang B, Situ H, Lin Y, Wang Z. XIAOPI Formula Inhibits Breast Cancer Stem Cells via Suppressing Tumor-Associated Macrophages/C-X-C Motif Chemokine Ligand 1 Pathway. Front Pharmacol. 2019 Nov 15;10:1371. doi: 10.3389/fphar.2019.01371. eCollection 2019. PMID 31803057
- [Background] Wang N, Yang B, Muhetaer G, Wang S, Zheng Y, Lu J, Li M, Zhang F, Situ H, Lin Y, Wang Z. XIAOPI formula promotes breast cancer chemosensitivity via inhibiting CXCL1/HMGB1-mediated autophagy. Biomed Pharmacother. 2019 Dec;120:109519. doi: 10.1016/j.biopha.2019.109519. Epub 2019 Oct 17. PMID 31629951
- [Background] Zheng Y, Wang N, Wang S, Yang B, Situ H, Zhong L, Lin Y, Wang Z. XIAOPI formula inhibits the pre-metastatic niche formation in breast cancer via suppressing TAMs/CXCL1 signaling. Cell Commun Signal. 2020 Mar 26;18(1):48. doi: 10.1186/s12964-020-0520-6. PMID 32213179